CLINICAL TRIAL: NCT00939263
Title: Development, Validation and Evaluation of an Adult and Pediatric Eosinophilic Esophagitis Activity Index: A Prospective Multicenter Study
Brief Title: Development, Validation and Evaluation of an Adult and Pediatric Eosinophilic Esophagitis Activity Index
Acronym: EEsAI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Bern (Other); Kantonsspital Olten (Other); Luzerner Kantonsspital (Other); Mayo Clinic (Other); University of Cincinnati (Other); University of Colorado, Denver (Other); Northwestern University (Other); Indiana University School of Medicine (Other); Philadelphia University (Other)
Responsible Party: Sponsor
Other Study IDs: 231/08; 0901 (Other: Ethikkommision KiKli BE)
Record Dates: First submitted 2009-07-13; First posted 2009-07-14 (Estimated); Last update posted 2015-09-16 (Estimated); Status verified 2015-09

CONDITIONS: Deglutition Disorders; Esophageal Diseases; Eosinophilia
Keywords: deglutition disorders; esophageal diseases; eosinophilia
MeSH Terms: conditions — Deglutition Disorders; Esophageal Diseases; Eosinophilia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: cohorts 1 (item weighting phase): 100 children with Eosinophilic Esophagitis, 150 adults with Eosinophilic Esophagitis
  Interventions: Other: assessment of disease activity using the EEsAI
- 2: cohorts 2 (evaluation phase): 200 children with Eosinophilic Esophagitis, 200 adults with Eosinophilic Esophagitis
  Interventions: Other: assessment of disease activity using the EEsAI

INTERVENTIONS:
Other: assessment of disease activity using the EEsAI — disease activity index

SUMMARY:
Eosinophilic Esophagitis (EoE) is a chronic inflammatory disease of the esophagus affecting children and adults. The most frequent symptoms are swallowing difficulties and thoracic pain. The disease has first been described in the 1980s and is found with rapidly increasing frequency mainly in industrialized countries. The factors that lead to EoE are until now incompletely understood, of importance, the disease is found more frequently in men and patients suffering from allergic diseases (e.g., Asthma). So far there exists no activity index to define the severity of EoE; such an index is urgently needed for future clinical trials to determine the efficacy of current and future therapies. The investigators' 3-year project, carried out in cooperation with international EoE experts, aims at the development of an activity index for adult and pediatric EoE patients that will be used in future clinical trials as well as observational studies.

DETAILED DESCRIPTION:
Background:

1. Introduction Coordinated by the Swiss Eosinophilic Esophagitis Research Group and in close collaboration with The International Gastrointestinal Eosinophil Researchers (TIGERS), we plan to conduct a series of related studies in order to develop an Activity Index (AI) for adult and pediatric patients with Eosinophilic Esophagitis (EoE).

EoE is an emerging disease, with rapidly growing clinical relevance and research activities. A validated assessment instrument is therefore urgently needed.

The purpose of this project is to develop within a representative group of pediatric and adult EoE-experienced gastroenterologists and EoE-experienced pathologists an AI for this chronic inflammatory esophageal disease. The project is investigator initiated, but funding from different sources will be necessary. The project will be conducted in compliance with this protocol, with the ICH guideline E6 on Good Clinical Practice, the FDA perspectives on patient-reported outcomes to support medical product labeling claims (1,2), and the applicable regulatory requirements.

As EoE is a new disorder we include below a comprehensive description of the disease.

1.1. Characterization of Eosinophilic Esophagitis Definition: EoE is rapidly emerging as a distinctive disorder in pediatric and adult gastroenterology. EoE is a chronic-inflammatory esophageal disease, characterized clinicopathologically by the presence of esophagus-related symptoms and by a dense esophageal eosinophilia, both of which persist despite prolonged treatment with proton pump inhibitors (3). Epidemiology: EoE is diagnosed 2-3 times more frequently in males than in females.

The disease is found mainly in industrialized countries such as the United States, Canada, Europe and Australia. EoE is likely to be a 'young' disease: it had not been seen prior to the early 1980, and there is strong evidence to suggest that its prevalence is increasing (4)(5). A population-based study performed in Switzerland suggested an increase in prevalence from 2 per 100000 to 40 per 100000 inhabitants over a 19-year period (6). Clinical Symptoms: As in many other diseases, symptom presentation differs significantly between children and adults. In infants and toddlers, food refusal is a common symptom of EoE. Children often suffer from GERD-like symptoms, vomiting and abdominal pain. Dysphagia and food impaction are reported increasingly with proceeding age. Adolescents and adults present mostly with dysphagia for solids and food impaction (5-7). Endoscopy/Histology: Esophago-gastro-duodenoscopy (EGD) is the first diagnostic step in the evaluation of an individual with suspected EoE. A broad spectrum of endoscopic features associated with EoE have been described, but the endoscopic suspicion needs confirmation by histology. The key diagnostic criterion for diagnosing EoE is an increased number of intraepithelial eosinophils in patients with lack of responsiveness to high-dose proton pump inhibition or normal pH-monitoring of the distal esophagus. In a consensus conference a cut-off value of =15 Eos/HPF (peak eosinophilic count in 400 fold magnification) in any biopsy was recommended as diagnostic criterion (3). Treatment: The optimal treatment for EoE is not yet clear, as experience has been limited largely to case series and small controlled trials. So far topically and systemically administered corticosteroids, several types of allergen-reduced diets, immunosuppressants and IL-5 blocking agents have been shown to be efficacious (8-11).

1.2. Rationale for the planned Studies In the clinical setting the current status of a given disease is often reported as "mild", "moderate" and "severe", and the course of the disease over time is described with terms such as "stable", "progressive", "in remission" or "flare-up". None of these terms has so far been clearly defined for EoE. However, an increasing number of phase 3 therapeutic multi-center trials and natural history studies in patients with EoE will be performed in the near future. In order to set up standardized study protocols and to compare results between different studies a standardized definition of disease activity is a necessity. Taken together, for clinical and for research purposes it is indispensable to define the terms mentioned above by a suitable, reproducible and validated score, which reflects the disease activity as precisely as possible. The necessity for such a score has repeatedly been discussed by the TIGERS and has been underscored by several publications (12).

Objective

The planned research program has the aim to develop and validate an AI for EoE (EEsAI) for adult (adEEsAI) and pediatric (pedEEsAI) patients, which can be used in future clinical trials and observational studies. According to the characterization of EoE, the AI will likely contain clinical and histopathological items. Laboratory and endoscopical parameters may be part of the score, but in a subsidiary role.

Methods:

The development and validation of a disease activity index is a research program involving several related studies. Broadly speaking, it involves 3 main steps: Step I Item Generation and Reduction through a Delphi process with an international expert group (Development phase A). Step II Item Weighting and Activity Index Derivation, using data from a first cohort of adult and a first cohort of pediatric patients (Development phase B).

Step III Evaluation of the Activity Index using data from a second independent cohort of adult and pediatric patients respectively. This involves also assessment of test-retest reliability and responsiveness of the score, using longitudinal data from the same patients.

ELIGIBILITY:
Inclusion Criteria:

* every patient with the diagnosis Eosinophilic Esophagitis
* pediatric and adult EoE patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult and pediatric patients with the diagnosis Eosinophilic Esophagitis, who are treated in the participating hospitals
Sampling Method: Non-Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2011-01; Primary Completion 2016-07 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Development of an EE Activity Index | 12 months

SECONDARY OUTCOMES:
Evaluation and validation of the activity index | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Alain Schoepfer, MD, PD+MER1, Principal Investigator — Department of Gastroenterology and Hepatology, Centre Hospitalier Universitaire Vaudois / CHUV; Alex Straumann, MD, Prof., Study Chair — Praxis Römerhof, Olten, Switzerland; Marcel Zwahlen, PhD, Prof., Study Director — Institute for Social and Preventive Medicine, University of Bern; Claudia Kuehni, MD MSc, Prof., Study Director — Institute for Social and Preventive Medicine, University of Bern; Christian Bussmann, MD, Study Director — Viollier AG
Locations (25):
- United States (14):
  - Gastroenterology and Hepatology : Mayo Clinic, Scottsdale, Scottsdale, Arizona
  - Department of Pediatrics : University of California, San Diego, California
  - The Children's Hospital : University of Colorado Denver, Aurora, Colorado
  - Gastroenterology and Hepatology : Mayo Clinic, Jacksonville, Jacksonville, Florida
  - Division of Gastroenterology : Northwestern University Chicago, Chicago, Illinois
  - Gastroenterology, hepatology and nutrition : Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Riley Hospital for Children : Indiana University School of Medicine, Indianapolis, Indiana
  - Institute for Clinical Research and Health Policy Studies: Tufts Medical Center, Boston, Massachusetts
  - Division of Allergy and Inflammation : Harvard Medical School Boston, Brookline, Massachusetts
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Pediatrics : Mount Sinai School of Medicine, New York, New York
  - Gastroenterology, Hepatology and Nutrition : University of Cincinnati, Cincinnati, Ohio
  - Children's Hospital of Philadelphia : University of Philadelphia, Philadelphia, Pennsylvania
  - Inova Fairfax Hospital for Children, Fairfax, Virginia
- Canada (2):
  - Clinical Epidemiology & Biostatistics : Mc Master University, Hamilton, Ontario
  - Ste-Justine Hospital : University of Montreal, Montreal, Quebec
- Switzerland (8):
  - Department of Gastroenterology, Inselspital/Bern University Hospital, Bern
  - Pädiatrische Gastroenterologie Medizinische Universitäts-Kinderklinik Bern, Bern
  - Institute for Social and Preventive Medicine, University of Bern, Bern
  - University Hospital Lausanne (CHUV), Lausanne
  - Department of Gastroenterology and Hepatology, Kantonsspital Lucerne, Lucerne
  - Institute for Pathology, Kantonsspital Lucerne, Lucerne
  - Praxis Römerhof, Römerstr. 7, Olten, Olten
  - Ostschweizer Kinderspital, Sankt Gallen
- Northumbria Healthcare Foundation Trust North Tyneside Hospital, North Shields, United Kingdom

REFERENCES:
- [Background] U.S. Department of Health and Human Services FDA Center for Drug Evaluation and Research; U.S. Department of Health and Human Services FDA Center for Biologics Evaluation and Research; U.S. Department of Health and Human Services FDA Center for Devices and Radiological Health. Guidance for industry: patient-reported outcome measures: use in medical product development to support labeling claims: draft guidance. Health Qual Life Outcomes. 2006 Oct 11;4:79. doi: 10.1186/1477-7525-4-79. PMID 17034633
- [Background] Patrick DL, Burke LB, Powers JH, Scott JA, Rock EP, Dawisha S, O'Neill R, Kennedy DL. Patient-reported outcomes to support medical product labeling claims: FDA perspective. Value Health. 2007 Nov-Dec;10 Suppl 2:S125-37. doi: 10.1111/j.1524-4733.2007.00275.x. PMID 17995471
- [Background] Furuta GT, Liacouras CA, Collins MH, Gupta SK, Justinich C, Putnam PE, Bonis P, Hassall E, Straumann A, Rothenberg ME; First International Gastrointestinal Eosinophil Research Symposium (FIGERS) Subcommittees. Eosinophilic esophagitis in children and adults: a systematic review and consensus recommendations for diagnosis and treatment. Gastroenterology. 2007 Oct;133(4):1342-63. doi: 10.1053/j.gastro.2007.08.017. Epub 2007 Aug 8. PMID 17919504
- [Background] Straumann A, Simon HU. Eosinophilic esophagitis: escalating epidemiology? J Allergy Clin Immunol. 2005 Feb;115(2):418-9. doi: 10.1016/j.jaci.2004.11.006. No abstract available. PMID 15696105
- [Background] Noel RJ, Putnam PE, Rothenberg ME. Eosinophilic esophagitis. N Engl J Med. 2004 Aug 26;351(9):940-1. doi: 10.1056/NEJM200408263510924. No abstract available. PMID 15329438
- [Background] Straumann A, Spichtin HP, Grize L, Bucher KA, Beglinger C, Simon HU. Natural history of primary eosinophilic esophagitis: a follow-up of 30 adult patients for up to 11.5 years. Gastroenterology. 2003 Dec;125(6):1660-9. doi: 10.1053/j.gastro.2003.09.024. PMID 14724818
- [Background] Liacouras CA, Spergel JM, Ruchelli E, Verma R, Mascarenhas M, Semeao E, Flick J, Kelly J, Brown-Whitehorn T, Mamula P, Markowitz JE. Eosinophilic esophagitis: a 10-year experience in 381 children. Clin Gastroenterol Hepatol. 2005 Dec;3(12):1198-206. doi: 10.1016/s1542-3565(05)00885-2. PMID 16361045
- [Background] Guyatt GH, Deyo RA, Charlson M, Levine MN, Mitchell A. Responsiveness and validity in health status measurement: a clarification. J Clin Epidemiol. 1989;42(5):403-8. doi: 10.1016/0895-4356(89)90128-5. PMID 2659745
- [Derived] Schoepfer AM, Hirano I, Coslovsky M, Roumet MC, Zwahlen M, Kuehni CE, Hafner D, Alexander JA, Dellon ES, Gonsalves N, Leung J, Bussmann C, Collins MH, Newbury RO, Smyrk TC, Woosley JT, Yang GY, Romero Y, Katzka DA, Furuta GT, Gupta SK, Aceves SS, Chehade M, Spergel JM, Falk GW, Meltzer BA, Comer GM, Straumann A, Safroneeva E; International EEsAI Study Group. Variation in Endoscopic Activity Assessment and Endoscopy Score Validation in Adults With Eosinophilic Esophagitis. Clin Gastroenterol Hepatol. 2019 Jul;17(8):1477-1488.e10. doi: 10.1016/j.cgh.2018.11.032. Epub 2018 Nov 23. PMID 30476587
- [Derived] Safroneeva E, Straumann A, Coslovsky M, Zwahlen M, Kuehni CE, Panczak R, Haas NA, Alexander JA, Dellon ES, Gonsalves N, Hirano I, Leung J, Bussmann C, Collins MH, Newbury RO, De Petris G, Smyrk TC, Woosley JT, Yan P, Yang GY, Romero Y, Katzka DA, Furuta GT, Gupta SK, Aceves SS, Chehade M, Spergel JM, Schoepfer AM; International Eosinophilic Esophagitis Activity Index Study Group. Symptoms Have Modest Accuracy in Detecting Endoscopic and Histologic Remission in Adults With Eosinophilic Esophagitis. Gastroenterology. 2016 Mar;150(3):581-590.e4. doi: 10.1053/j.gastro.2015.11.004. Epub 2015 Nov 14. PMID 26584601
- [Derived] Safroneeva E, Coslovsky M, Kuehni CE, Zwahlen M, Haas NA, Panczak R, Taft TH, Hirano I, Dellon ES, Gonsalves N, Leung J, Bussmann C, Woosley JT, Yan P, Romero Y, Furuta GT, Gupta SK, Aceves SS, Chehade M, Straumann A, Schoepfer AM; International EEsAI Study Group. Eosinophilic oesophagitis: relationship of quality of life with clinical, endoscopic and histological activity. Aliment Pharmacol Ther. 2015 Oct;42(8):1000-10. doi: 10.1111/apt.13370. Epub 2015 Aug 14. PMID 26271642
- [Derived] Schoepfer AM, Straumann A, Panczak R, Coslovsky M, Kuehni CE, Maurer E, Haas NA, Romero Y, Hirano I, Alexander JA, Gonsalves N, Furuta GT, Dellon ES, Leung J, Collins MH, Bussmann C, Netzer P, Gupta SK, Aceves SS, Chehade M, Moawad FJ, Enders FT, Yost KJ, Taft TH, Kern E, Zwahlen M, Safroneeva E; International Eosinophilic Esophagitis Activity Index Study Group. Development and validation of a symptom-based activity index for adults with eosinophilic esophagitis. Gastroenterology. 2014 Dec;147(6):1255-66.e21. doi: 10.1053/j.gastro.2014.08.028. Epub 2014 Aug 23. PMID 25160980